CLINICAL TRIAL: NCT03347279
Title: A Multicentre, Randomized, Double-Blind, Placebo Controlled, Parallel Group, Phase 3 Study to Evaluate the Efficacy and Safety of Tezepelumab in Adults and Adolescents With Severe Uncontrolled Asthma (NAVIGATOR)
Brief Title: Study to Evaluate Tezepelumab in Adults & Adolescents With Severe Uncontrolled Asthma
Acronym: NAVIGATOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5180C00007
Record Dates: First submitted 2017-11-09; First posted 2017-11-20 (Actual); Results first posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-10

CONDITIONS: Asthma
Keywords: Asthma, Uncontrolled Asthma, Severe Uncontrolled Asthma
MeSH Terms: conditions — Asthma | interventions — tezepelumab

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 1:1 ratio to either tezepelumab or matching placebo both administered subcutaneously.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tezepelumab (Experimental): Tezepelumab: Tezepelumab subcutaneous injection
  Interventions: Biological: Experimental: Tezepelumab
- Placebo (Placebo Comparator): Placebo: Placebo subcutaneous injection
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Experimental: Tezepelumab — Tezepelumab subcutaneous injection
  Other Names: Tezepelumab
  Arms: Tezepelumab
Other: Placebo — Placebo subcutaneous injection
  Arms: Placebo

SUMMARY:
A Multicentre, Randomized, Double-Blind, Placebo Controlled, Parallel Group, Phase 3 Study to Evaluate the Efficacy and Safety of Tezepelumab in Adults and Adolescents with Severe Uncontrolled Asthma

DETAILED DESCRIPTION:
This is a multicentre, randomized, double-blind, placebo controlled, parallel group study designed to evaluate the efficacy and safety of tezepelumab in adults and adolescents with severe, uncontrolled asthma on medium to high-dose ICS and at least one additional asthma controller medication with or without OCS. Approximately 1060 subjects will be randomized globally. Subjects will receive tezepelumab, or placebo, administered via subcutaneous injection at the study site, over a 52-week treatment period. The study also includes a post-treatment follow-up period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age. 12-80
* Documented physician-diagnosed asthma for at least 12 months
* Subjects who have received a physician-prescribed asthma controller medication with medium or high dose ICS for at least 12 months.
* Documented treatment with a total daily dose of either medium or high dose ICS (≥ 500 µg fluticasone propionate dry powder formulation equivalent total daily dose) for at least 3 months.
* At least one additional maintenance asthma controller medication is required according to standard practice of care and must be documented for at least 3 months.
* Morning pre-BD FEV1 <80% predicted normal (<90% for subjects 12-17 yrs)
* Evidence of asthma as documented by either: Documented historical reversibility of FEV1 ≥12% and ≥200 mL in the previous 12 months OR Post-BD (albuterol/salbutamol) reversibility of FEV1 ≥12% and ≥200 mL during screening.
* Documented history of at least 2 asthma exacerbation events within 12 months.
* ACQ-6 score ≥1.5 at screening and on day of randomization

Exclusion Criteria:

* Pulmonary disease other than asthma.
* History of cancer.
* History of a clinically significant infection.
* Current smokers or subjects with smoking history ≥10 pack-years and subjects using vaping products, including electronic cigarettes.
* History of chronic alcohol or drug abuse within 12 months.
* Hepatitis B, C or HIV.
* Pregnant or breastfeeding.
* History of anaphylaxis following any biologic therapy.
* Subject randomized in the current study or previous tezepelumab studies.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1061 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2020-09-08 (Actual); Study Completion 2020-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Menzies-Gow, MD, Principal Investigator — Royal Brompton Hospital, United Kingdom
Locations (226):
- United States (82):
  - Research Site, Dothan, Alabama
  - Research Site, Foley, Alabama
  - Research Site, Gilbert, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Bakersfield, California
  - Research Site, Encinitas, California
  - Research Site, Huntington Beach, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Mission Viejo, California
  - Research Site, Newport Beach, California
  - Research Site, Northridge, California
  - Research Site, Palm Desert, California
  - Research Site, Rolling Hills Estates, California
  - Research Site, Walnut Creek, California
  - Research Site, Westminster, California
  - Research Site, Denver, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Celebration, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Orlando, Florida
  - Research Site, Panama City, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Sebring, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Fayetteville, Georgia
  - Research Site, Gainesville, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Stockbridge, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Michigan City, Indiana
  - Research Site, Fort Mitchell, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Lake Charles, Louisiana
  - Research Site, Zachary, Louisiana
  - Research Site, White Marsh, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Fall River, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Flint, Michigan
  - Research Site, Novi, Michigan
  - Research Site, Port Huron, Michigan
  - Research Site, Troy, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Northfield, New Jersey
  - Research Site, Toms River, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Valhalla, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Gastonia, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Mayfield Heights, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Edmond, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Warwick, Rhode Island
  - Research Site, Anderson, South Carolina
  - Research Site, Columbia, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Allen, Texas
  - Research Site, Amarillo, Texas
  - Research Site, Boerne, Texas
  - Research Site, Dallas, Texas
  - Research Site, Lampasas, Texas
  - Research Site, McAllen, Texas
  - Research Site, Plano, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Manassas, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Cudahy, Wisconsin
  - Research Site, Madison, Wisconsin
- Argentina (7):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, Mendoza
  - Research Site, Nueve de Julio
  - Research Site, Quilmes
- Australia (8):
  - Research Site, Campbelltown
  - Research Site, Kent Town
  - Research Site, Melbourne
  - Research Site, Nedlands
  - Research Site, New Lambton
  - Research Site, Spearwood
  - Research Site, Westmead
  - Research Site, Woolloongabba
- Austria (4):
  - Research Site, Klagenfurt
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Vienna
- Brazil (10):
  - Research Site, Blumenau
  - Research Site, Botucatu
  - Research Site, Curitiba
  - Research Site, Porto Alegre
  - Research Site, Recife
  - Research Site, Salvador
  - Research Site, Santo André
  - Research Site, São Bernardo do Campo
  - Research Site, Sorocaba
  - Research Site, Vitória
- Canada (12):
  - Research Site, Calgary, Alberta
  - Research Site, Sherwood Park, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Ajax, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Trois-Rivières, Quebec
- France (12):
  - Research Site, Brest
  - Research Site, Grenoble
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Strasbourg
  - Research Site, Toulouse
- Germany (10):
  - Research Site, Bamberg
  - Research Site, Berlin
  - Research Site, Frankfurt
  - Research Site, Frankfurt am Main
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Landsberg
  - Research Site, Leipzig
  - Research Site, Lübeck
  - Research Site, Mainz
- Israel (5):
  - Research Site, Ashkelon
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Rehovot
- Japan (39):
  - Research Site, Bunkyō City
  - Research Site, Chūōku
  - Research Site, Edogawa-ku
  - Research Site, Fujieda-shi
  - Research Site, Fukuoka
  - Research Site, Habikino-shi
  - Research Site, Hamamatsu
  - Research Site, Higashiibaraki-gun
  - Research Site, Himeji-shi
  - Research Site, Hitachi-shi
  - Research Site, Itabashi-ku
  - Research Site, Kagoshima
  - Research Site, Kanazawa
  - Research Site, Kasuga-shi
  - Research Site, Kishiwada-shi
  - Research Site, Kitakyushu
  - Research Site, Koga-shi
  - Research Site, Matsusaka-shi
  - Research Site, Meguro-ku
  - Research Site, Minatoku
  - Research Site, Mizunami-shi
  - Research Site, Nagaoka-shi
  - Research Site, Niigata
  - Research Site, Ogaki-shi
  - Research Site, Ohota-ku
  - Research Site, Omuta-shi
  - Research Site, Sagamihara-shi
  - Research Site, Sapporo
  - Research Site, Setagaya-ku
  - Research Site, Shibuya-ku
  - Research Site, Shinagawa-ku
  - Research Site, Shinjuku-ku
  - Research Site, Sumida-ku
  - Research Site, Takamatsu
  - Research Site, Toshima-ku
  - Research Site, Ube
  - Research Site, Yokkaichi-shi
  - Research Site, Yokohama
  - Research Site, Yoshida-gun
- Russia (3):
  - Research Site, Izhevsk
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Research Site, Jeddah, Saudi Arabia
- South Africa (12):
  - Research Site, Bellville
  - Research Site, Boksburg North
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, eMkhomazi
  - Research Site, Johannesburg
  - Research Site, Lenasia Ext8
  - Research Site, Middelburg
  - Research Site, Mowbray
  - Research Site, Parow
  - Research Site, Pretoria
  - Research Site, Witbank
- South Korea (8):
  - Research Site, Bucheon-si
  - Research Site, Cheongju-si
  - Research Site, Daegu
  - Research Site, Jeju City
  - Research Site, Jeonju
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suwon
- Taiwan (7):
  - Research Site, Hsinchu
  - Research Site, Kaohsiung City
  - Research Site, Kaohsiung Hsien
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Yilan
- Ukraine (2):
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv Region
- Research Site, London, United Kingdom
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Feleszko W, Caminati M, Gern JE, Johnston SL, Marchese C, Clarke D, Ambrose CS, Lindsley AW. Effect of tezepelumab on asthma exacerbations co-occurring with infection-attributed acute respiratory illnesses. Ann Allergy Asthma Immunol. 2026 Jan;136(1):61-65.e1. doi: 10.1016/j.anai.2025.09.015. Epub 2025 Oct 8. PMID 41072729
- [Derived] Yang X, Wang L, Huang K, Tang W, Berame EJ, Park HS, Hunter G, Jiang W, Wu CC, Min CW, Domek-Zielinska K, Lal H, Molfino NA, Ponnarambil SS, Zhong N. Efficacy and Safety of Tezepelumab in Adults With Severe, Uncontrolled Asthma in Asia: Results From the Phase 3 DIRECTION Study. J Allergy Clin Immunol Pract. 2025 Nov;13(11):3011-3020.e9. doi: 10.1016/j.jaip.2025.07.046. Epub 2025 Aug 7. PMID 40782846
- [Derived] Pavord ID, Brightling CE, Korn S, Martin NL, Ponnarambil SS, Molfino NA, Parnes JR, Ambrose CS. Tezepelumab can Restore Normal Lung Function in Patients with Severe, Uncontrolled Asthma: Pooled Results from the PATHWAY and NAVIGATOR Studies. Pulm Ther. 2025 Jun;11(2):315-325. doi: 10.1007/s41030-025-00294-2. Epub 2025 Apr 26. PMID 40285963
- [Derived] Jacobs JS, Han JK, Lee JK, Laidlaw TM, Martin NL, Caveney S, Ambrose CS, Martin N, Spahn JD, Hoyte FCL. Effect of Tezepelumab on Sino-Nasal Outcome Test (SNOT)-22 Domain and Symptom-Specific Scores in Patients with Severe, Uncontrolled Asthma and a History of Chronic Rhinosinusitis with Nasal Polyps. Adv Ther. 2025 Jan;42(1):510-522. doi: 10.1007/s12325-024-03006-5. Epub 2024 Nov 8. PMID 39514041
- [Derived] Wechsler ME, Brusselle G, Virchow JC, Bourdin A, Kostikas K, Llanos JP, Roseti SL, Ambrose CS, Hunter G, Jackson DJ, Castro M, Lugogo N, Pavord ID, Martin N, Brightling CE. Clinical response and on-treatment clinical remission with tezepelumab in a broad population of patients with severe, uncontrolled asthma: results over 2 years from the NAVIGATOR and DESTINATION studies. Eur Respir J. 2024 Dec 5;64(6):2400316. doi: 10.1183/13993003.00316-2024. Print 2024 Dec. PMID 39326921
- [Derived] Carr TF, Moore WC, Kraft M, Brusselle G, Castro M, Chupp GL, Wechsler ME, Hunter G, Lindsley AW, Llanos JP, Burke LK, Chandarana S, Ambrose CS. Efficacy of Tezepelumab in Patients with Severe, Uncontrolled Asthma Across Multiple Clinically Relevant Subgroups in the NAVIGATOR Study. Adv Ther. 2024 Jul;41(7):2978-2990. doi: 10.1007/s12325-024-02889-8. Epub 2024 May 27. PMID 38802635
- [Derived] Corren J, Menzies-Gow A, Bimmel J, McGuinness A, Almqvist G, Bowen K, Griffiths JM, Ponnarambil S, Bourdin A, Israel E, Colice G, Brightling CE, Wechsler ME; PATHWAY and NAVIGATOR study investigators. Tezepelumab for the treatment of severe asthma: a plain language summary of the PATHWAY and NAVIGATOR studies. Immunotherapy. 2023 Nov;15(16):1327-1340. doi: 10.2217/imt-2023-0109. Epub 2023 Sep 29. PMID 37772607
- [Derived] Menzies-Gow A, Ambrose CS, Colice G, Hunter G, Cook B, Molfino NA, Llanos JP, Israel E. Effect of Tezepelumab on Lung Function in Patients With Severe, Uncontrolled Asthma in the Phase 3 NAVIGATOR Study. Adv Ther. 2023 Nov;40(11):4957-4971. doi: 10.1007/s12325-023-02659-y. Epub 2023 Sep 19. PMID 37723356
- [Derived] Pavord ID, Hoyte FCL, Lindsley AW, Ambrose CS, Spahn JD, Roseti SL, Cook B, Griffiths JM, Hellqvist A, Martin N, Llanos JP, Martin N, Colice G, Corren J. Tezepelumab reduces exacerbations across all seasons in patients with severe, uncontrolled asthma (NAVIGATOR). Ann Allergy Asthma Immunol. 2023 Nov;131(5):587-597.e3. doi: 10.1016/j.anai.2023.08.015. Epub 2023 Aug 23. PMID 37619779
- [Derived] Menzies-Gow A, Bourdin A, Chupp G, Israel E, Hellqvist A, Hunter G, Roseti SL, Ambrose CS, Llanos JP, Cook B, Corren J, Colice G. Effect of tezepelumab on healthcare utilization in patients with severe, uncontrolled asthma: The NAVIGATOR study. Ann Allergy Asthma Immunol. 2023 Sep;131(3):343-348.e2. doi: 10.1016/j.anai.2023.05.028. Epub 2023 May 30. PMID 37263380
- [Derived] Corren J, Menzies-Gow A, Chupp G, Israel E, Korn S, Cook B, Ambrose CS, Hellqvist A, Roseti SL, Molfino NA, Llanos JP, Martin N, Bowen K, Griffiths JM, Parnes JR, Colice G. Efficacy of Tezepelumab in Severe, Uncontrolled Asthma: Pooled Analysis of the PATHWAY and NAVIGATOR Clinical Trials. Am J Respir Crit Care Med. 2023 Jul 1;208(1):13-24. doi: 10.1164/rccm.202210-2005OC. PMID 37015033
- [Derived] Menzies-Gow A, Wechsler ME, Brightling CE, Korn S, Corren J, Israel E, Chupp G, Bednarczyk A, Ponnarambil S, Caveney S, Almqvist G, Golabek M, Simonsson L, Lawson K, Bowen K, Colice G; DESTINATION study investigators. Long-term safety and efficacy of tezepelumab in people with severe, uncontrolled asthma (DESTINATION): a randomised, placebo-controlled extension study. Lancet Respir Med. 2023 May;11(5):425-438. doi: 10.1016/S2213-2600(22)00492-1. Epub 2023 Jan 23. PMID 36702146
- [Derived] Yin Z, Zhou Y, Turnquist HR, Liu Q. Neuro-epithelial-ILC2 crosstalk in barrier tissues. Trends Immunol. 2022 Nov;43(11):901-916. doi: 10.1016/j.it.2022.09.006. Epub 2022 Oct 14. PMID 36253275
- [Derived] Menzies-Gow A, Corren J, Bourdin A, Chupp G, Israel E, Wechsler ME, Brightling CE, Griffiths JM, Hellqvist A, Bowen K, Kaur P, Almqvist G, Ponnarambil S, Colice G. Tezepelumab in Adults and Adolescents with Severe, Uncontrolled Asthma. N Engl J Med. 2021 May 13;384(19):1800-1809. doi: 10.1056/NEJMoa2034975. PMID 33979488
- [Derived] Menzies-Gow A, Colice G, Griffiths JM, Almqvist G, Ponnarambil S, Kaur P, Ruberto G, Bowen K, Hellqvist A, Mo M, Garcia Gil E. NAVIGATOR: a phase 3 multicentre, randomized, double-blind, placebo-controlled, parallel-group trial to evaluate the efficacy and safety of tezepelumab in adults and adolescents with severe, uncontrolled asthma. Respir Res. 2020 Oct 13;21(1):266. doi: 10.1186/s12931-020-01526-6. PMID 33050934
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5180C00007&attachmentIdentifier=103f6433-96f8-44c4-b837-d7315e83136d&fileName=d5180c00007-csp-v5-14.May.2020_Redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5180C00007&attachmentIdentifier=3d32e500-6365-408d-bdb5-c145f83f1d2b&fileName=d5180c00007-sap-ed-4_22.Oct.2020_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1061 subjects were randomised at 231 centres in 17 countries to receive treatment with tezepelumab 210mg Q4W or placebo,
Pre-assignment Details: Of the 1061 randomised, 1059 (99.8%) subjects received treatment. 82 (7.7%) of the subjects randomised and treated were adolescents.
Groups:
- Tezepelumab 210mg Q4W: Tezepelumab administered every 4 weeks subcutaneously
- Placebo: Placebo administered subcutaneously
Period: Overall Study
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Started | 529 | 532
Received Treatment | 528 | 531
Completed | 513 | 509
Not Completed | 16 | 23
Not completed — Withdrawal by Subject | 8 | 15
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 5 | 2
Not completed — Did not receive treatment / Non-compliance with protocol / did not complete safety follow-up visits | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tezepelumab 210mg Q4W | Placebo | Total
Number analyzed (Participants) | 528 | 531 | 1059
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 41 | 41 | 82
  Between 18 and 65 years | 391 | 416 | 807
  >=65 years | 96 | 74 | 170
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.9 (16.3) | 49.0 (15.9) | 49.5 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 335 | 337 | 672
  Male | 193 | 194 | 387
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 332 | 327 | 659
  Black of African American | 30 | 31 | 61
  Asian | 146 | 149 | 295
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  American Indian or Alaska Native | 0 | 1 | 1
  Other | 19 | 23 | 42
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 83 | 81 | 164
  Not Hispanic or Latino | 445 | 450 | 895

OUTCOME MEASURES:

1. Primary Outcome: Annual Asthma Exacerbation Rate in Adult and Adolescent Patients With Uncontrolled Asthma
Description: The annual exacerbation rate is based on unadjudicated exacerbations reported by the investigator in the eCRF. The analysis is based on the primary population (Full Analysis Set)
Time Frame: From randomisation to Study Week 52.
Measure: Least Squares Mean (95% Confidence Interval); unit: events per year
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 528 | 531
events per year | 0.93 [0.80 to 1.07] | 2.10 [1.84 to 2.39]
Statistical Analysis 1: Comparison: Tezepelumab 210mg Q4W vs Placebo; Test type: Superiority; p < 0.001, Negative Binomial; Rate Ratio = 0.44, 95% CI 2-sided [0.37 to 0.53]

2. Primary Outcome: Annual Asthma Exacerbation Rate in Adult and Adolescent Patients With Uncontrolled Asthma in Subjects With Baseline Eosinophils < 300 Cells/uL
Description: The annual exacerbation rate is based on unadjudicated exacerbations reported by the investigator in the eCRF. This analysis is based on subjects with baseline eosinophils < 300 cells/uL
Time Frame: From randomisation to Study Week 52.
Measure: Least Squares Mean (95% Confidence Interval); unit: events per year
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 309 | 309
events per year | 1.02 [0.84 to 1.23] | 1.73 [1.46 to 2.05]
Statistical Analysis 1: Comparison: Tezepelumab 210mg Q4W vs Placebo; Test type: Superiority; p < 0.001, Negative Binomial; Rate Ratio = 0.59, 95% CI 2-sided [0.46 to 0.75]

3. Secondary Outcome: Mean Change From Baseline at Week 52 in Pre-dose/Pre-bronchodilator (Pre-BD) Forced Expiratory Volume in 1 Second (FEV1) (L) (Key Secondary Endpoint)
Description: Mean change from baseline in FEV1 as compared to placebo at Week 52. FEV1 is defined as the volume of air exhaled from the lungs in the first second of a forced expiration.
Time Frame: From randomisation to Study Week 52
Population: Number of participants analyzed is the number of subjects with an observation at Week 52. All subjects from the Full Analysis Set with at least one change from baseline value at any post baseline visit contributes to the analyses.
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 471 | 453
Litre | 0.23 (0.018) | 0.10 (0.018)
Statistical Analysis 1: Comparison: Tezepelumab 210mg Q4W vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Least Squares (LS) Mean Difference = 0.13, 95% CI 2-sided [0.08 to 0.18]

4. Secondary Outcome: Mean Change From Baseline at Week 52 in Standardized Asthma Quality of Life Questionnaire for 12 Years and Older (AQLQ(S)+12) Total Score (Key Secondary Endpoint)
Description: Mean change from baseline in AQLQ(S)+12 as compared to placebo at Week 52. The AQLQ(S)+12 is a questionnaire that measures the health-related quality of life experienced by asthma subjects. The total score is defined as the average of all 32 questions in the AQLQ(S)+12 questionnaire. AQLQ(S)+12 is a 7-point scale questionnaire, ranging from 7 (no impairment) to 1 (severe impairment).
Time Frame: From randomisation to Study Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Scale of score
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 480 | 467
Scale of score | 1.48 (0.049) | 1.14 (0.049)
Statistical Analysis 1: Comparison: Tezepelumab 210mg Q4W vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Means Difference = 0.33, 95% CI 2-sided [0.2 to 0.47]

5. Secondary Outcome: Mean Change From Baseline at Week 52 in Asthma Control Questionnaire-6(ACQ-6) (Key Secondary Endpoint)
Description: Change from baseline in ACQ-6 as compared to placebo at Week 52. The ACQ-6 captures asthma symptoms and short-acting β2-agonist use via subject-report. Questions are weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The ACQ-6 score is the mean of the responses.
Time Frame: From randomisation to Study Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Scale of score
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 485 | 472
Scale of score | -1.53 (0.045) | -1.20 (0.046)
Statistical Analysis 1: Comparison: Tezepelumab 210mg Q4W vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Means Difference = -0.33, 95% CI 2-sided [-0.46 to -0.2]

6. Secondary Outcome: Mean Change From Baseline at Week 52 in Asthma Symptom Diary (Key Secondary Endpoint)
Description: Mean change from baseline at Week 52 in Asthma Symptom Diary. The Asthma Symptom Diary comprises of 10 items (5 items in the morning; 5 items in the evening). Asthma symptoms during night time and daytime are recorded by the patient each morning and evening in the daily diary. A daily ASD score is the mean of the 10 items. Responses for all 10 items are required to calculate the daily ASD score; otherwise, it is treated as missing. For the 7-day average asthma symptom score, scoring is done with no imputation using the mean of at least 4 of the 7 daily ASD scores as a mean weekly item score. The 7-day average ASD score ranges from 0 to 4, where 0 indicates no asthma symptoms.
Time Frame: From randomisation to Study Week 52
Population: Number of participants analyzed is the number of subjects with a weekly mean at Week 52. All subjects from the Full Analysis Set with at least one change from baseline weekly mean at any post-baseline week contributes to the analyses.
Measure: Least Squares Mean (Standard Error); unit: Scale of score
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 374 | 355
Scale of score | -0.70 (0.027) | -0.59 (0.027)
Statistical Analysis 1: Comparison: Tezepelumab 210mg Q4W vs Placebo; Test type: Superiority; p = 0.004, Mixed Models Analysis; LS Means Difference = -0.11, 95% CI 2-sided [-0.19 to -0.04]

7. Secondary Outcome: Time to First Asthma Exacerbation
Description: Time to first occurrence of asthma exacerbation post-randomisation, presented as number of subjects with at least one asthma exacerbation as reported by the investigator in the eCRF.
Time Frame: From randomisation to Study Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 528 | 531
Participants | 231 | 319

8. Secondary Outcome: Mean Change From Baseline at Week 52 in Clinic Fractional Exhaled Nitric Oxide (FeNO) (Ppb)
Description: Mean change from baseline at Study Week 52 in FeNO (ppb) measured at site
Time Frame: From randomisation to Study Week 52
Measure: Least Squares Mean (Standard Error); unit: ppb
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 440 | 426
ppb | -17.29 (1.156) | -3.46 (1.165)

9. Secondary Outcome: Mean Change From Baseline in Daily Rescue Medication Use (Weekly Means) at Week 52
Description: Daily rescue medication use is defined as: Number of night inhaler puffs + 2 x [number of night nebulizer times] + number of daytime inhaler puffs + 2 x [number of day nebulizer times]. Weekly means are calculated using at least 4 of 7 days of daily rescue medication use.
Time Frame: From randomisation to Study Week 52
Measure: Least Squares Mean (Standard Error); unit: weekly mean rescue medication use
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 439 | 428
weekly mean rescue medication use | -2.53 (0.137) | -2.36 (0.137)

10. Secondary Outcome: Mean Change From Baseline in Work Productivity Loss Due to Asthma at Week 52
Description: WPAI+CIQ (Work Productivity and Activity Impairment plus Classroom Impairment Questionnaire) contains 10 questions. Work productivity loss is derived by sum of percentage of missed work due to asthma and product of percentage of actual working hours times degree of asthma affecting work productivity while working. Percentage of missed work due to asthma is calculated by number of hours missed work due to asthma divided by total number of hours missed work plus number of hours actually worked.
Time Frame: From randomisation to Study Week 52
Population: The work productivity loss is only applicable to subjects who were employed, which is a subset of the study population.
Measure: Mean (Standard Deviation); unit: Percentage of work productivity loss
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 185 | 177
Percentage of work productivity loss | -20.16 (30.31) | -16.58 (29.46)

11. Secondary Outcome: Mean Change From Baseline in Class Productivity Loss Due to Asthma at Week 52
Description: WPAI+CIQ (Work Productivity and Activity Impairment plus Classroom Impairment Questionnaire) contains 10 questions. Class productivity loss is derived by sum of percentage of missed class hours due to asthma and product of percentage of actual hours in class times degree of asthma affecting productivity while in class. Percentage of missed hours in class due to asthma is calculated by number of hours in class missed due to asthma divided by total number of hours in class missed plus number of hours actually in class.
Time Frame: From randomisation to Study Week 52
Population: The class productivity loss is only applicable to subjects attending school, which is a subset of the study population.
Measure: Mean (Standard Deviation); unit: Percentage of class productivity loss
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 15 | 19
Percentage of class productivity loss | -14.03 (33.00) | -24.72 (26.48)

12. Secondary Outcome: Activity Impairment at Week 52
Description: WPAI+CIQ (Work Productivity and Activity Impairment plus Classroom Impairment Questionnaire) contains 10 questions. Activity impairment is the degree health affected regular activities (other than work or class) rated from 0 to 10, with 0 meaning no effect, divided by 10, and then expressed as a percentage.
Time Frame: From randomisation to Study Week 52
Measure: Mean (Standard Deviation); unit: Percentage of activity impairment
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 401 | 393
Percentage of activity impairment | -20.0 (28.6) | -17.9 (27.1)

13. Secondary Outcome: Pharmacokinetics of Tezepelumab
Description: Mean serum trough PK concentrations taken pre-dose at each visit
Time Frame: Pre-dose samples at Baseline, Week 4, Week 12, Week 24, Week 36, Week 52, Week 64
Population: Number of subjects who received at least one dose of IP. Number analysed at each timepoint is a subset of this based on subjects who had sample results available at that timepoint. The placebo arm is not applicable since it is not the experimental product.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 528 | 0
ug/mL
  Baseline: number analyzed (Participants) | 524 | 0
  Baseline | 0 (0) |
  Week 4: number analyzed (Participants) | 514 | 0
  Week 4 | 10.1573 (74.51) |
  Week 12: number analyzed (Participants) | 491 | 0
  Week 12 | 18.7396 (48.53) |
  Week 24: number analyzed (Participants) | 461 | 0
  Week 24 | 20.1924 (51.77) |
  Week 36: number analyzed (Participants) | 464 | 0
  Week 36 | 19.5246 (55.58) |
  Week 52: number analyzed (Participants) | 452 | 0
  Week 52 | 19.8894 (70.04) |
  Week 64: number analyzed (Participants) | 72 | 0
  Week 64 | 1.7675 (171.86) |

14. Secondary Outcome: Mean Change From Baseline at Week 52 in EQ-5D-5L VAS
Description: Mean change from baseline at Study Week 52 in EQ-5D-5L VAS. EQ-5D-5L visual analogue scale (VAS) allows subjects to rate current health status on a scale of 0-100, with 0 being the worst imaginable health state.
Time Frame: At Study Week 52
Measure: Least Squares Mean (Standard Error); unit: scale of score
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 448 | 435
scale of score | 14.64 (0.708) | 11.86 (0.712)

15. Secondary Outcome: Clinicians Global Impression of Change at Week 52
Description: CGIC (Clinical global impression of change) is an overall evaluation of response to treatment, conducted by investigator using 7-point rating scale, ranging from 1 (very much improved), to 7 (very much worse)
Time Frame: From randomisation to Study Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 483 | 477
Participants
  Very much improved | 96 | 60
  Much improved | 199 | 132
  Minimally improved | 98 | 131
  No change | 77 | 130
  Minimally worse | 11 | 19
  Much worse | 2 | 4
  Very much worse | 0 | 1

16. Secondary Outcome: Patients Global Impression of Change at Week 52
Description: PGIC (Patient global impression of change) is an overall evaluation of response to treatment, conducted by the patient using 7-point rating scale, ranging from 1 (very much improved), to 7 (very much worse).
Time Frame: From randomisation to Study Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 479 | 466
Participants
  Very much improved | 255 | 182
  Much Improved | 103 | 94
  Minimally improved | 71 | 76
  No change | 39 | 99
  Minimally worse | 6 | 8
  Much worse | 4 | 6
  Very much worse | 1 | 1

17. Secondary Outcome: Patients Global Impression of Severity at Week 52
Description: PGI-S (Patient global impression of severity) is an overall evaluation of patient's perception of overall symptom severity using a 6-point rating scale, ranging from 0 = No symptoms, 1=Very mild symptoms, 2=Mild symptoms, 3=Moderate symptoms, 4=Severe symptoms, 5=Very severe symptoms
Time Frame: At Study Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 479 | 466
Participants
  No symptoms | 118 | 78
  Very mild symptoms | 138 | 128
  Mild symptoms | 110 | 128
  Moderate symptoms | 99 | 111
  Severe symptoms | 14 | 19
  Very severe symptoms | 0 | 2

18. Secondary Outcome: Mean Change From Baseline at Week 52 in Blood Eosinophils (Cells/uL)
Description: Mean change from baseline at Study Week 52 in blood eosinophils (cells/uL)
Time Frame: From randomisation to Study Week 52
Measure: Least Squares Mean (Standard Error); unit: cells/uL
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 458 | 451
cells/uL | -170.02 (9.222) | -40.15 (9.254)

19. Secondary Outcome: Mean Change From Baseline at Week 52 in Total Serum IgE (IU/mL)
Description: Mean change from baseline at Study Week 52 in total serum IgE (IU/mL)
Time Frame: From randomisation to Study Week 52
Measure: Least Squares Mean (Standard Error); unit: IU/mL
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 482 | 471
IU/mL | -164.38 (34.414) | 43.61 (34.542)

20. Secondary Outcome: Number of Participants With Asthma Specific Healthcare Utilization Over 52 Weeks
Description: Number of participants with asthma specific healthcare utilizations (e.g. unscheduled physician visits, unscheduled phone calls to physicians, use of other asthma medications) over 52 weeks
Time Frame: From randomisation to Study Week 52
Measure: Number; unit: Participants
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 528 | 531
Participants
  Hospitalisation | 17 | 37
  Emergency Room visit | 23 | 50
  Unscheduled visit to specialist | 187 | 231
  Home visit | 9 | 10
  Telephone call | 101 | 133
  Ambulance transport | 4 | 12

21. Secondary Outcome: Mean Change From Baseline in Home Based Morning Peak Expiratory Flow (PEF) at Week 52 (Weekly Means)
Description: Mean change from baseline in home based morning PEF (L/min) at Study Week 52. Home PEF testing will be performed by the subject in the morning upon awakening and in the evening at bedtime using an electronic, hand-held spirometer. Weekly means are calculated using at least 4 of the 7 days of PEF data.
Time Frame: From randomisation to Study Week 52
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 414 | 391
L/min | 34.57 (3.051) | 18.01 (3.074)

22. Secondary Outcome: Mean Change From Baseline in Home Based Evening Peak Expiratory Flow (PEF) at Week 52 (Weekly Means)
Description: Mean change from baseline in home based evening PEF (L/min) at Study Week 52. Home PEF testing will be performed by the subject in the morning upon awakening and in the evening at bedtime using an electronic, hand-held spirometer. Weekly means are calculated using at least 4 of the 7 days of PEF data.
Time Frame: From randomisation to Study Week 52
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 405 | 390
L/min | 23.87 (3.075) | 9.01 (3.094)

23. Secondary Outcome: Mean Change From Baseline in Night Time Awakenings (Weekly Means) at Week 52
Description: Mean change from baseline in night time awakenings due to asthma at Study Week 52. Night-time awakenings percentage defined as number of nights with awakenings due to asthma and requiring rescue medication divided by number of nights with data and multiplied by 100%. At least 4 out of 7 days of data is required to calculate a weekly mean.
Time Frame: From randomisation to Study Week 52
Measure: Least Squares Mean (Standard Error); unit: percentage of nights with awakenings
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 418 | 395
percentage of nights with awakenings | -33.51 (1.381) | -30.22 (1.387)

24. Secondary Outcome: Immunogenecity of Tezepelumab
Description: Anti-drug antibodies (ADA) responses at baseline and post baseline. Persistently positive is defined as positive at >=2 post baseline assessments (with >=16 weeks between the first and the last positive) or positive at last post baseline assessment. Transiently positive is defined as having at least one post baseline ADA positive assessment and not fulfilling the conditions of persistently positive. Treatment boosted ADA defined as baseline positive ADA that was boosted to a 4 fold or higher level following treatment. Treatment emergent ADA defined as sum of treatment induced ADA and treatment boosted ADA.
Time Frame: Baseline, and from time of first dose at Week 0 to end of study at Week 64.
Measure: Number; unit: Participants
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 527 | 530
Participants
  ADA positive at baseline and/or post-baseline | 26 | 44
  Any baseline ADA positive | 17 | 25
  Only baseline ADA positive | 14 | 8
  Any post-baseline ADA positive | 12 | 36
  Both baseline and >= 1 post-baseline ADA positive | 3 | 17
  Treatment induced ADA positive | 9 | 18
  Treatment boosted ADA positive | 1 | 2
  Treatment emergent ADA positive | 10 | 20
  ADA persistently positive | 4 | 18
  ADA transiently positive | 8 | 18

25. Secondary Outcome: Proportion of Subjects Who Had no Asthma Exacerbations
Description: The proportion of subjects who have no exacerbations is presented as the percentage of subjects with no exacerbations. This is defined as subjects who meet both the following criteria: (1) completed the 52 week treatment period and (2) did not report an exacerbation during this period.
Time Frame: From randomisation to Study Week 52
Measure: Number; unit: Percentage
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 528 | 531
Percentage | 54.2 | 38.6

26. Secondary Outcome: Annual Asthma Exacerbation Rate Resulting in Emergency Room Visit or Hospitalisation
Description: The annualized exacerbation rate is based on exacerbations reported by the investigator that are associated with an emergency room visit, urgent care visit, or a hospitalization (where urgent care visit was captured as an emergency room visit on the eCRF)
Time Frame: From randomisation to Study Week 52
Measure: Least Squares Mean (95% Confidence Interval); unit: events per year
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 528 | 531
events per year | 0.06 [0.04 to 0.09] | 0.28 [0.20 to 0.39]

27. Secondary Outcome: Proportion of Subjects With at Least One Asthma Exacerbation Associated With Emergency Room Visit or Hospitalisation
Description: Proportion of subjects with at least one asthma exacerbation associated with emergency room visit or hospitalisation as recorded by the investigator in the CRF. This is presented as percentage of subjects with at least one asthma exacerbation associated with emergency room visit or hospitalisation.
Time Frame: From randomisation to Study Week 52
Measure: Number; unit: Percentage
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 528 | 531
Percentage | 4.7 | 12.2

28. Secondary Outcome: Proportion of Subjects Who Had no Asthma Exacerbations Associated With Emergency Room or Hospitalisation
Description: The proportion of subjects with no exacerbations is presented as percentage of subjects who meet both the following criteria: (1) completed the 52 week treatment period and (2) did not report an exacerbation associated with emergency room or hospitalisation during this period.
Time Frame: From randomisation to Study Week 52
Measure: Number; unit: Percentage
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 528 | 531
Percentage | 92.4 | 85.1

29. Other Pre Specified Outcome: Annual Asthma Exacerbation Rate Associated With Hospitalisations
Description: The annualized exacerbation rate is based on exacerbations reported by the investigator that are associated with hospitalization
Time Frame: From randomisation to Study Week 52
Measure: Least Squares Mean (95% Confidence Interval); unit: events per year
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 528 | 531
events per year | 0.03 [0.01 to 0.06] | 0.19 [0.12 to 0.30]

30. Other Pre Specified Outcome: Annual Asthma Exacerbation Rate Using Adjudicated Data
Description: The annualized exacerbation rate is based on exacerbations as defined for the primary endpoint, but any hospitalisation and ER visits which are adjudicated to be asthma related are added, and those adjudicated to not be asthma related are removed from analyses.
Time Frame: From randomisation to Study Week 52
Measure: Least Squares Mean (95% Confidence Interval); unit: events per year
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 528 | 531
events per year | 0.94 [0.81 to 1.09] | 2.14 [1.88 to 2.44]

31. Other Pre Specified Outcome: Annual Asthma Exacerbation Rate Associated With Emergency Room (ER) Visit or Hospitalisation Using Adjudicated Data
Description: The annualized exacerbation rate is based on exacerbations associated with hospitalisations or ER visits, where hospitalisation and ER visits adjudicated to be asthma related are added, and those adjudicated to not be asthma related are removed from analyses.
Time Frame: From randomisation to Study Week 52
Measure: Least Squares Mean (95% Confidence Interval); unit: events per year
Arm/Group | Tezepelumab 210mg Q4W | Placebo
Number analyzed (Participants) | 528 | 531
events per year | 0.08 [0.05 to 0.12] | 0.31 [0.22 to 0.42]

ADVERSE EVENTS:
Time Frame: From first dose of study drug until end of study at Week 64.
Arm/Group | Tezepelumab 210mg Q4W | Placebo
All-Cause Mortality (participants affected / at risk) | 0/528 | 2/531
Serious Adverse Events (participants affected / at risk) | 52/528 | 73/531
Other Adverse Events (participants affected / at risk) | 306/528 | 331/531
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tezepelumab 210mg Q4W (N=528) | Placebo (N=531)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (2) | 1 (1)
Uveitis (Eye disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (2)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal achalasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (3)
Pancreatitis necrotising (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Breast abscess (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster oticus (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 2 (4)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 2 (2)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bone cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cubital tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Idiopathic generalised epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (2)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 14 (15) | 39 (81)
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cyanosis (Vascular disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tezepelumab 210mg Q4W (N=528) | Placebo (N=531)
Bronchitis bacterial (Infections and infestations) | 24 (26) | 17 (20)
Urinary tract infection (Infections and infestations) | 22 (33) | 22 (24)
Viral upper respiratory tract infection (Infections and infestations) | 17 (21) | 13 (18)
Influenza like illness (General disorders) | 19 (21) | 22 (26)
Bronchitis (Infections and infestations) | 25 (39) | 33 (36)
Gastroenteritis (Infections and infestations) | 17 (18) | 14 (15)
Nasopharyngitis (Infections and infestations) | 113 (172) | 114 (188)
Pharyngitis (Infections and infestations) | 17 (18) | 15 (17)
Rhinitis (Infections and infestations) | 14 (18) | 17 (37)
Sinusitis (Infections and infestations) | 19 (22) | 40 (56)
Upper respiratory tract infection (Infections and infestations) | 58 (94) | 88 (129)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (25) | 13 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 21 (26) | 15 (16)
Headache (Nervous system disorders) | 43 (96) | 45 (68)
Asthma (Respiratory, thoracic and mediastinal disorders) | 14 (17) | 23 (25)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 16 (19) | 17 (25)
Hypertension (Vascular disorders) | 23 (27) | 22 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/79/NCT03347279/Prot_002.pdf
  • Statistical Analysis Plan (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/79/NCT03347279/SAP_003.pdf